CLINICAL TRIAL: NCT04409990
Title: Shear Wave Elastography of Rectal Adenomas and Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SWE of rectal lesions
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Rectal Neoplasms; Elasticity Imaging Techniques
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shear Wave Elastography (Other): SWE value measurement will be added during the ERUS examination.
  Interventions: Diagnostic Test: Shear Wave Elastography

INTERVENTIONS:
Diagnostic Test: Shear Wave Elastography — SWE value of rectal lesions

SUMMARY:
The diagnosis of rectal lesions is a challenging task, and the accuracy of the primary staging is important preoperatively. A relatively novel technology makes it possible to measure the tissue stiffness during endorectal ultrasonography.

The purpose of this study is to evaluate the diagnostic value of Shear Wave Elastography (SWE). The hypothesis is that the tissue stiffness is higher in malignant tissue than in benign lesions.

DETAILED DESCRIPTION:
This study will include patients with an endoscopy verified rectal lesion referred to the radiology department for pretreatment evaluation.

During the investigation, patients will undergo magnetic resonance imaging (MRI) and endorectal ultrasonography (ERUS). During the ERUS, the tissue stiffness of the lesion and visible lymph nodes will be measured using the SWE technology.

Hypotheses:

1. Tumour stiffness measurement by SWE gives a statistically significantly higher value in malignant processes than in benign rectal tumors.
2. Tissue stiffness measurement with SWE gives a statistically significantly higher value in lymph node metastases than in reactive enlarged lymph nodes.
3. There is a statistically significant correlation between SWE and MRI apparent diffusion coefficient (ADC)

Histopathology report of surgical specimen will serve as endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Adults above 18 years of age
* Rectal lesions discovered during endoscopy
* Lesions located no more than 15 cm above the anal verge

Exclusion Criteria:

* Non-eligibility for MRI (e.g. claustrophobia, implants)
* Preoperative radiotherapy and/or chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
SWE accuracy | 1 month
  The accuracy of SWE value as compared with the histopathology report

SECONDARY OUTCOMES:
SWE and ADC measurement | 1 week
  The correlation between ERUS SWE and MRI ADC value

CONTACTS AND LOCATIONS:
Overall Officials: Søren R Rafaelsen, DMSc, Study Chair — Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li T, Lu M, Li Y, Li J, Hu Z, Li X, Cheng X, Jiang J, Tan B. Quantitative Elastography of Rectal Lesions: The Value ofShear Wave Elastography in Identifying Benign and Malignant Rectal Lesions. Ultrasound Med Biol. 2019 Jan;45(1):85-92. doi: 10.1016/j.ultrasmedbio.2018.09.008. Epub 2018 Oct 17. PMID 30342780